CLINICAL TRIAL: NCT07297524
Title: A Single-Center, Single-Arm Exploratory Study to Evaluate the Impact of Multimodal Acoustic Therapy (MAT) on Objective and Subjective Auditory Perception During a 12-Week Intervention and a 12-Week Follow-Up in Pediatric and Adolescent Cochlear Implant Users
Brief Title: CRESCENDO: ChildREn's muSiC ENhancement in Cochlear Implant Users
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: BELL Therapeutics Inc. (Industry)
Responsible Party: Principal Investigator, Sang-Yeon Lee, Assistant Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2404-090-1531
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cochlear Implant; Hearing Loss
Keywords: Multimodal Acoustic Therapy; Cochlear Implant; Pediatric Cochlear Implant Users; Adolescent Cochlear Implant Users; Auditory Rehabilitation; Mobile Application; Digital Health Intervention
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Device: Auditory rehabilitation application Application: Wowfit
  Interventions: Device: Mobile Auditory Rehabilitation

INTERVENTIONS:
Device: Mobile Auditory Rehabilitation — Mobile Application for Auditory Rehabilitation

SUMMARY:
This exploratory, single-center, single-arm study investigates the impact of a 12-week Multimodal Acoustic Therapy (MAT) intervention followed by a 12-week follow-up period on both objective and subjective auditory perception in pediatric cochlear implant users.

DETAILED DESCRIPTION:
Duration of study period (per participant): 24 weeks, including a 12-week intervention and a 12-week online follow-up.

Participants will use the Multimodal Acoustic Therapy (MAT) mobile application at home for 12 weeks to improve music and speech perception.

Participants will visit the site twice (baseline and post-intervention), while all other evaluations, including follow-up, will be conducted online.

The first on-site visit is mainly to on-board participants and to train them for accurate use of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with cochlear implants
* Korean patients aged 10 to 19 years
* Capable of using a smartphone
* Scored ≤80% on MCI pre-assessment
* Voluntarily agreed to participate in this study

Exclusion Criteria:

* Has systemic medical conditions (e.g., cancer, stroke) that limit daily functioning
* Has intellectual disability, congenital malformation, or other neurological disorders affecting language or cognitive abilities
* Has diagnosed emotional disorders such as depression or anxiety
* Primarily uses sign language for daily communication
* Has undergone cochlear implant revision surgery
* Has prior experience with the investigational auditory rehabilitation application used in this study

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Melody Contour Identification (MCI) | 12 weeks
  Participants complete a melody contour identification task in which they listen to brief melodic sequences and select the contour pattern (e.g., rising, falling, flat).
  Performance is quantified as the percentage of correctly identified contours (% correct).
  Higher scores indicate better melody contour perception.

SECONDARY OUTCOMES:
Music-Related Quality of Life (MuRQoL) | 12 weeks
  Each item is rated on a 1-5 Likert scale, and domain scores may be converted to a normalized 0-100 scale.
  Higher scores indicate better music-related quality of life.
Parents' Evaluation of Aural/Oral Performance of Children (PEACH) | 12 weeks
  Auditory performance in everyday listening situations will be evaluated using the Parents' Evaluation of Aural/Oral Performance of Children (PEACH) questionnaire.
  Parents rate their child's functional auditory behaviors across quiet and noisy environments.
  Scores are converted to a percentage (0-100%), with higher scores indicating better auditory performance.
  The PEACH is a parent-proxy assessment tool, consistent with its standard scoring procedure.
Quality of Life - Cochlear Implants (Parent-Proxy Report) | 12 weeks
  Quality of life specific to pediatric cochlear implant users will be assessed using the Quality of Life - Cochlear Implants (CI-QOL) questionnaire.
  This is a parent-proxy reported measure, in which parents rate their child's auditory-related daily functioning, communication abilities, social participation, and emotional well-being.
  Scores range from 0 to 100, with higher scores indicating better quality of life.
Emotional Prosody Perception Test (EPP) | 12 weeks
  Performance will be reported as the percentage. Higher percentages indicate better emotional prosody perception.
Monosyllabic Word Test | 4 weeks
  Performance will be reported as the percentage of correctly identified words (% correct).
  Higher percentages indicate better auditory word recognition ability.
Sentence Test in Quiet | 4 weeks
  Performance will be reported as the percentage of correctly repeated sentences (% correct).
  Higher percentages indicate better speech recognition ability.
Speech test in Noise | 4 weeks
  Sentence recognition will be assessed using standardized sentence materials presented in background noise at a +5 dB signal-to-noise ratio (SNR), where the noise level is higher relative to the speech signal.
  Performance will be reported as the percentage of correctly repeated sentences (% correct).
  Lower percentages are expected compared to quiet due to increased listening difficulty; higher percentages indicate better speech-in-noise perception ability.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea